CLINICAL TRIAL: NCT03026712
Title: Association of Dual Transcranial Electrical Stimulation (tDCS) to Upper Limb Robotic Therapy in Individuals With Chronic Stroke
Brief Title: Hemiparetic Arm Robotic Mobilization With Non Invasive Electrical Stimulation
Acronym: hARMonies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Giovanni Morone, MD, PhD, MD, PhD, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FSLCBM01
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Stroke; Paresis; Upper Extremity Paralysis
Keywords: Robotic therapy; tDCS; non invasive electrical stimulation; ArmeoPower; interhemispheric balance
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real tDCS (Experimental)
  Interventions: Device: Real dual tDCS + Robotic Arm Therapy
- Sham tDCS (Sham Comparator)
  Interventions: Device: SHAM tDCS + Robotic Arm Therapy

INTERVENTIONS:
Device: Real dual tDCS + Robotic Arm Therapy — Dual tDCS (anodic on injured hemisphere, cathodic on healthy hemisphere). Motor cortex will be simultaneously stimulated at an intensity equal to 1-2 mA and for a maximum duration of 20 minutes just before 30 minutes of arm robotic task oriented treatment performed with an exoskeleton device (Armeo Power).
  The intervention will be performed 5 times per week for 2 consecutive weeks.
  Arms: Real tDCS
Device: SHAM tDCS + Robotic Arm Therapy — SHAM bilateral tDCS for a maximum duration of 20 minutes just before 30 minutes of arm robotic task oriented treatment performed with an exoskeleton device (Armeo Power).
  The intervention will be performed 5 times per week for 2 consecutive weeks.
  Arms: Sham tDCS

SUMMARY:
The two cerebral hemispheres find themselves in a state of balanced mutual inhibition. A stroke with involvement of motor function leads to a reduced excitability in affected hemisphere M1 and to an increased excitability of contralateral M1. Stroke therefore might impair interhemispheric balance, leading to a decreased inhibition of contralesional hemisphere by ipsilesional hemisphere and, in turn, to an increased inhibition of ipsilesional hemisphere by contralesional hemisphere. Permanence of healthy hemisphere hyperactivation in chronic phase after stroke is usually index of little functional recovery and is correlated with a greater ipsilateral structural damage.

Robot-mediated physical therapy is an innovative rehabilitation technique that is effective in stroke patients. In this study, the investigators will add a non-invasive brain stimulation protocol with Transcranial stimulation with direct current (tDCS) to the robotic treatment in chronic stroke patients. tDCS is a non-invasive brain stimulation technique that is able to modulate cortical excitability. The hypothesis is that dual t-DCS (ipsilesional excitation and concomitant contralesional inhibition) could restore interhemispheric balance improving the benefits of robotic therapy with Armeo Power®.

DETAILED DESCRIPTION:
The general theory of the inhibitory interhemispheric competition speculates that, under physiological conditions, the two cerebral hemispheres find themselves in a state of balanced mutual inhibition. Accordingly, some electrophysiological and functional imaging studies have shown that a stroke with involvement of motor function leads to a reduced excitability in affected hemisphere M1 and to an increased excitability of contralateral M1. Stroke therefore might impair interhemispheric balance, leading to a decreased inhibition of contralesional hemisphere by ipsilesional hemisphere and, in turn, to an increased inhibition of ipsilesional hemisphere by contralesional hemisphere.

This imbalance in cerebral hemispheres excitability tends to decline over the functional recovery in the first months after stroke, in proportion to the functional recovery of the ipsilateral structures.

Alternatively, permanence of healthy hemisphere hyperactivation in chronic phase after stroke is usually index of little functional recovery and is correlated with a greater structural damage to the ipsilesional corticospinal tract and transcallosal fibers, although some studies have suggested a vicarious role of healthy hemisphere.

Recently, some authors have proposed a structural reserve-based bimodal model of recovery, for which the vicarious model would be valid only for patients with poor structural reserves (and therefore more extensive damage), while the interhemispheric competition model would be valid for patients with larger structural reserves.

In the light of these data, it is conceivable that procedures aiming at promoting the re-establishment of a normal balance in interhemispheric interaction can facilitate motor function recovery of the paretic limb, at least in patients with appropriate structural reserves.

Transcranial stimulation with direct current (tDCS) is a non-invasive brain stimulation technique that uses low intensity electrical current at constant voltage and variable duration that is able to modulate cortical excitability efficiently, lastingly (with effects that begin during stimulation and that last for a few hours from the end of the stimulation) and safely in healthy subjects: moreover, it is able to produce changes of excitability in both directions (i.e. towards an increase and towards its reduction) in dependence of electrodes positioning on the scalp.

Specifically, t-DCS appears to induce metaplasticity phenomena, that is a polarity-dependent modulation of the response to subsequent synaptic potentiation protocols. Considering these results and the conclusions of a recent meta-analysis, it seems appropriate to expose a patient to t-DCS immediately before or in the early stage of intervention aiming at promoting synaptic plasticity, such as neuro-rehabilitation techniques.

Alongside the traditional physical therapy techniques, during the last twenty years many research groups around the world have started to develop robots supporting physical treatments.

A review on robot-mediated physical therapy clinical trials shows how this innovative rehabilitation technique is effective both in acute and chronic stroke patients, although it is not proven its superiority over traditional rehabilitation methods.

In this study, the investigators will use a robotic exoskeleton that allows targeted interventions on specific tasks in the three spatial dimensions; this robot, marketed under the name Armeo Power® (Hocoma AG, Switzerland), is one of the most advanced rehabilitation devices for the upper limb. The effectiveness of this tool has been demonstrated in a recent multicenter trial of chronic stroke patients with moderate-severe upper limb motor deficit.

The purpose of this study is to evaluate the benefits arising from the combination of dual t-DCS (ipsilesional excitation and contralesional inhibition) and robotic therapy with Armeo Power® in the treatment of chronic stroke patients with upper limb paralysis.

This study is a double blind randomized controlled trial in which chronic stroke patients with upper limb paresis undergone robotic treatment with Armeo Power® will be randomized to concomitant dual tDCS (excitatory on injured side and inhibitory on health side) o sham tDCS.

All patients will undergo an initial evaluation before starting treatment (between 30 and 15 days before the start) where it will be filled in a form with the medical history and the personal data and will be signed informed consent.

Once eligible, the patient will be subjected to a first clinical evaluation using validated scales, a kinematic evaluation of upper limb motor performance with ArmeoPower® and a neurophysiological evaluation.

At the end of the evaluation, every patient will be assigned through a randomized system to one of two study groups:

* Group A: robotic treatment with Armeo Power® associated with REAL dual tDCS (anodic on injured hemisphere, cathodic on healthy hemisphere) - 40 patients
* Group B: robotic treatment with Armeo Power® associated with SHAM dual tDCS - 40 patients

Immediately prior the start of treatment (time T-1), every participant will perform a second clinical assessment and kinematic evaluation and will begin treatment on the same day in the gym of the Private Department of Saint Lucia Foundation.

The ArmeoPower® device is an exoskeleton robot for upper limb rehabilitation able to allow the patients' execution of movements of proximal (shoulder-elbow movements) and distal (movements of the wrist) segments of upper limb.

Once the arms of the robot are adapted to patent's upper limb, the exoskeleton is mounted and set for defining the action areas and the volumes of exploration.

At the beginning of each session, ArmeoPower® exoskeleton will be mounted according to the patients' stored settings, which takes about 10 minutes.

Once mounted, it will proceed to real or sham tDCS stimulation, depending on the group the patient belong to.

Participants in group A will perform real dual tDCS stimulation immediately before each session of the robotic treatment, while patients in group B will perform the treatment with robotics platform with the same intensity and duration of group A but preceded by sham dual tDCS stimulation.

Real dual tDCS stimulation requires the application of the anode over the injured motor cortex (M1) and of the cathode on the healthy motor cortex (M1), so as to simultaneously perform an excitability suppression of healthy hemisphere and an activation of the ischemic cortex.

Motor cortex will be simultaneously stimulated at an intensity equal to 1-2 mA and for a maximum duration of 20 minutes. Sham dual t-DCS requires the application of the electrodes in the same positions and for the same duration, but without the delivery of electrical stimulation.

The robotic rehabilitation treatment will be started immediately after the end of stimulation, and the actual treatment will last for 30 minutes. The robot is able to relieve the weight of the arm and assisting the patient during motor execution. The patient sees on a monitor the targets upon which he should move the effector and executes the movement through the active assistance of the robot, which compensates the patient's motor deficits. Videogame-based exercises and functional training exercises of daily life activities are carried out with visual, acoustic and performance feedback. A physical therapist with a specific training certificate is always present during the sessions, with 1:1 ratio with patients.

Each patient will perform 5 sessions per week for two consecutive weeks, after which will be performed clinical, kinematic and neurophysiological evaluations expected to T0; the patient will then be re-evaluated in follow-up at one month (T1) and at 3 months after the end of treatment (T2), with clinical and kinematic assessments.

Data will be analyzed using parametric statistics if will appear to be normally distributed (based on Kolgomorov-Smirnov test with Lilliefors correction), in particular by applying a two-way mixed model analysis of variance (with an intra- and inter-factor between subjects). If the data won't appear to be normally distributed, they will be analyzed using Friedman's analysis for the intra-subject variations, and by Mann-Whitney u-test for variations between the two groups. The level of significance will be set at 0.05 for all analysis, except for post-hoc to which is applied the Bonferroni correction.

Guidelines for the safe use of non-invasive brain stimulation (Wassermann, 1998) will be respected; the participants should be able to signed an informed consent.

There are not literature report of adverse events or contraindications with regard to the use of ArmeoPower® robotics platform, except for patients with severe deformities of the paretic upper limb, that are excluded from this study. Data on patients will be anonymous and stored with password protection. There will be no samples of biological material, drug delivery, healthy volunteers or animals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with isolated ischemic stroke, confirmed by brain imaging (MRI, CT)
* subjects who retain sufficient cognitive functions and language to follow the instructions given by doctors and therapists
* subjects with basal Modified Ashworth Scale score under 3
* subjects with basal Fugl-Meyer score ≥ 3 so that they are not completely paralyzed
* subjects who have signed informed consent to participate in this study
* subjects that show stable conditions in the two pre-treatment evaluations, in order to avoid "Hawthorne effect"

Exclusion Criteria:

* subjects with chronic paretic limb deformities
* subjects with complete and flaccid paralysis of all motor performances of shoulder and elbow;
* subjects with severe hemineglect (Pizzamiglio battery for unilateral spatial neglect including letter cancellation test, barrage tests, reading and Wundt-Jastro area illusion test; patients diagnosed with neglect if 3 of 4 items of this battery are present)
* subjects showing an increase in the Fugl-Meyer more than 2.1 points in the second pre-treatment clinical evaluation, compared to the score of the first evaluation
* subjects with contraindications to the execution of transcranial magnetic stimulation - TMS - (pacemakers, metal implants)
* subjects with epilepsy
* Previous neurosurgical interventions
* Severe upper limb osteoporosis
* Upper limb strength or joint movement limitation due to previous fractures
* Upper limb strength or joint movement limitation due to previous surgical interventions
* Mini Mental State Evaluation (MMSE) <24

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Significant Fugl-Meyer Assessment Upper Extremity (FMA-UE) improvement in real dual tDCS group vs sham tDCS group | first assessment will occur within 2 days from enrollment, and will be repeated within 2 days from the end of 2 week-training and at 1 and 3 months follow-up

SECONDARY OUTCOMES:
Significant Modified Ashworth scale improvement in real dual tDCS group vs sham tDCS group | first assessment will occur within 2 days from enrollment, and will be repeated within 2 days from the end of 2 week-training and at 1 and 3 months follow-up
Significant Action Research Arm Test (ARAT) improvement in real dual tDCS group vs sham tDCS group | first assessment will occur within 2 days from enrollment, and will be repeated within 2 days from the end of 2 week-training and at 1 and 3 months follow-up
Significant Barthel index improvement in real dual tDCS group vs sham tDCS group | first assessment will occur within 2 days from enrollment, and will be repeated within 2 days from the end of 2 week-training and at 1 and 3 months follow-up
Significant kinematic performance improvement, measured by ArmeoPower®, in real dual tDCS group vs sham tDCS group | first assessment will occur within 2 days from enrollment, and will be repeated within 2 days from the end of 2 week-training
Significant rebalancing of motor evoked potential (MEP) laterality index in real dual tDCS group vs sham tDCS group | first assessment will occur within 2 days from enrollment, and will be repeated within 2 days from the end of 2 week-training

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Paolucci, Study Director — I.R.C.C.S. Fondazione Santa Lucia, Roma; Vincenzo Di Lazzaro, Study Director — Policlinico Universitario Campus Bio-Medico, Roma
Locations (2):
- Italy (2):
  - I.R.C.C.S. Fondazione Santa Lucia, Rome
  - Policlinico Universitario Campus Bio-Medico, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chollet F, DiPiero V, Wise RJ, Brooks DJ, Dolan RJ, Frackowiak RS. The functional anatomy of motor recovery after stroke in humans: a study with positron emission tomography. Ann Neurol. 1991 Jan;29(1):63-71. doi: 10.1002/ana.410290112. PMID 1996881
- [Background] Cicinelli P, Traversa R, Rossini PM. Post-stroke reorganization of brain motor output to the hand: a 2-4 month follow-up with focal magnetic transcranial stimulation. Electroencephalogr Clin Neurophysiol. 1997 Dec;105(6):438-50. doi: 10.1016/s0924-980x(97)00052-0. PMID 9448645
- [Background] Kinsbourne, M. (1974). Mechanisms of hemispheric interaction in man. In Hemispheric Disconnection and Cerebral Function, M. Kinsbourne, and W. Smith, eds. (Springfield: Charles C Thomas).
- [Background] Cramer SC, Nelles G, Benson RR, Kaplan JD, Parker RA, Kwong KK, Kennedy DN, Finklestein SP, Rosen BR. A functional MRI study of subjects recovered from hemiparetic stroke. Stroke. 1997 Dec;28(12):2518-27. doi: 10.1161/01.str.28.12.2518. PMID 9412643
- [Background] Cunningham DA, Machado A, Janini D, Varnerin N, Bonnett C, Yue G, Jones S, Lowe M, Beall E, Sakaie K, Plow EB. Assessment of inter-hemispheric imbalance using imaging and noninvasive brain stimulation in patients with chronic stroke. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S94-103. doi: 10.1016/j.apmr.2014.07.419. Epub 2014 Sep 3. PMID 25194451
- [Background] Delvaux V, Alagona G, Gerard P, De Pasqua V, Pennisi G, de Noordhout AM. Post-stroke reorganization of hand motor area: a 1-year prospective follow-up with focal transcranial magnetic stimulation. Clin Neurophysiol. 2003 Jul;114(7):1217-25. doi: 10.1016/s1388-2457(03)00070-1. PMID 12842718
- [Background] Di Lazzaro V, Pilato F, Dileone M, Profice P, Capone F, Ranieri F, Musumeci G, Cianfoni A, Pasqualetti P, Tonali PA. Modulating cortical excitability in acute stroke: a repetitive TMS study. Clin Neurophysiol. 2008 Mar;119(3):715-723. doi: 10.1016/j.clinph.2007.11.049. Epub 2007 Dec 31. PMID 18165149
- [Background] Di Pino G, Pellegrino G, Assenza G, Capone F, Ferreri F, Formica D, Ranieri F, Tombini M, Ziemann U, Rothwell JC, Di Lazzaro V. Modulation of brain plasticity in stroke: a novel model for neurorehabilitation. Nat Rev Neurol. 2014 Oct;10(10):597-608. doi: 10.1038/nrneurol.2014.162. Epub 2014 Sep 9. PMID 25201238
- [Background] Duque J, Hummel F, Celnik P, Murase N, Mazzocchio R, Cohen LG. Transcallosal inhibition in chronic subcortical stroke. Neuroimage. 2005 Dec;28(4):940-6. doi: 10.1016/j.neuroimage.2005.06.033. Epub 2005 Aug 9. PMID 16084737
- [Background] Gerloff C, Bushara K, Sailer A, Wassermann EM, Chen R, Matsuoka T, Waldvogel D, Wittenberg GF, Ishii K, Cohen LG, Hallett M. Multimodal imaging of brain reorganization in motor areas of the contralesional hemisphere of well recovered patients after capsular stroke. Brain. 2006 Mar;129(Pt 3):791-808. doi: 10.1093/brain/awh713. Epub 2005 Dec 19. PMID 16364955
- [Background] Grefkes C, Fink GR. Connectivity-based approaches in stroke and recovery of function. Lancet Neurol. 2014 Feb;13(2):206-16. doi: 10.1016/S1474-4422(13)70264-3. PMID 24457190
- [Background] Hummel FC, Cohen LG. Non-invasive brain stimulation: a new strategy to improve neurorehabilitation after stroke? Lancet Neurol. 2006 Aug;5(8):708-12. doi: 10.1016/S1474-4422(06)70525-7. PMID 16857577
- [Background] Jang SH, Kwon HG. Change of the anterior corticospinal tract on the normal side of the brain in chronic stroke patients: Diffusion tensor imaging study. Somatosens Mot Res. 2015;32(1):25-30. doi: 10.3109/08990220.2014.949006. Epub 2014 Aug 28. PMID 25166214
- [Background] Jang SH, Kim K, Kim SH, Son SM, Jang WH, Kwon HG. The relation between motor function of stroke patients and diffusion tensor imaging findings for the corticospinal tract. Neurosci Lett. 2014 Jun 20;572:1-6. doi: 10.1016/j.neulet.2014.04.044. Epub 2014 May 4. PMID 24796808
- [Background] Kang N, Summers JJ, Cauraugh JH. Transcranial direct current stimulation facilitates motor learning post-stroke: a systematic review and meta-analysis. J Neurol Neurosurg Psychiatry. 2016 Apr;87(4):345-55. doi: 10.1136/jnnp-2015-311242. Epub 2015 Aug 28. PMID 26319437
- [Background] Klamroth-Marganska V, Blanco J, Campen K, Curt A, Dietz V, Ettlin T, Felder M, Fellinghauer B, Guidali M, Kollmar A, Luft A, Nef T, Schuster-Amft C, Stahel W, Riener R. Three-dimensional, task-specific robot therapy of the arm after stroke: a multicentre, parallel-group randomised trial. Lancet Neurol. 2014 Feb;13(2):159-66. doi: 10.1016/S1474-4422(13)70305-3. Epub 2013 Dec 30. PMID 24382580
- [Background] Liebetanz D, Nitsche MA, Tergau F, Paulus W. Pharmacological approach to the mechanisms of transcranial DC-stimulation-induced after-effects of human motor cortex excitability. Brain. 2002 Oct;125(Pt 10):2238-47. doi: 10.1093/brain/awf238. PMID 12244081
- [Background] Liepert J, Bauder H, Wolfgang HR, Miltner WH, Taub E, Weiller C. Treatment-induced cortical reorganization after stroke in humans. Stroke. 2000 Jun;31(6):1210-6. doi: 10.1161/01.str.31.6.1210. PMID 10835434
- [Background] Maraka S, Jiang Q, Jafari-Khouzani K, Li L, Malik S, Hamidian H, Zhang T, Lu M, Soltanian-Zadeh H, Chopp M, Mitsias PD. Degree of corticospinal tract damage correlates with motor function after stroke. Ann Clin Transl Neurol. 2014 Nov;1(11):891-9. doi: 10.1002/acn3.132. Epub 2014 Oct 31. PMID 25540803
- [Background] Murase N, Duque J, Mazzocchio R, Cohen LG. Influence of interhemispheric interactions on motor function in chronic stroke. Ann Neurol. 2004 Mar;55(3):400-9. doi: 10.1002/ana.10848. PMID 14991818
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Nitsche MA, Nitsche MS, Klein CC, Tergau F, Rothwell JC, Paulus W. Level of action of cathodal DC polarisation induced inhibition of the human motor cortex. Clin Neurophysiol. 2003 Apr;114(4):600-4. doi: 10.1016/s1388-2457(02)00412-1. PMID 12686268
- [Background] Prange GB, Jannink MJ, Groothuis-Oudshoorn CG, Hermens HJ, Ijzerman MJ. Systematic review of the effect of robot-aided therapy on recovery of the hemiparetic arm after stroke. J Rehabil Res Dev. 2006 Mar-Apr;43(2):171-84. doi: 10.1682/jrrd.2005.04.0076. PMID 16847784
- [Background] Ranieri F, Podda MV, Riccardi E, Frisullo G, Dileone M, Profice P, Pilato F, Di Lazzaro V, Grassi C. Modulation of LTP at rat hippocampal CA3-CA1 synapses by direct current stimulation. J Neurophysiol. 2012 Apr;107(7):1868-80. doi: 10.1152/jn.00319.2011. Epub 2012 Jan 11. PMID 22236710
- [Background] Rosso C, Valabregue R, Attal Y, Vargas P, Gaudron M, Baronnet F, Bertasi E, Humbert F, Peskine A, Perlbarg V, Benali H, Lehericy S, Samson Y. Contribution of corticospinal tract and functional connectivity in hand motor impairment after stroke. PLoS One. 2013 Sep 27;8(9):e73164. doi: 10.1371/journal.pone.0073164. eCollection 2013. PMID 24086272
- [Background] Schulz R, Braass H, Liuzzi G, Hoerniss V, Lechner P, Gerloff C, Hummel FC. White matter integrity of premotor-motor connections is associated with motor output in chronic stroke patients. Neuroimage Clin. 2014 Nov 18;7:82-6. doi: 10.1016/j.nicl.2014.11.006. eCollection 2015. PMID 25610769
- [Background] Schulz R, Frey BM, Koch P, Zimerman M, Bonstrup M, Feldheim J, Timmermann JE, Schon G, Cheng B, Thomalla G, Gerloff C, Hummel FC. Cortico-Cerebellar Structural Connectivity Is Related to Residual Motor Output in Chronic Stroke. Cereb Cortex. 2017 Jan 1;27(1):635-645. doi: 10.1093/cercor/bhv251. PMID 26508336
- [Background] Schulz R, Koch P, Zimerman M, Wessel M, Bonstrup M, Thomalla G, Cheng B, Gerloff C, Hummel FC. Parietofrontal motor pathways and their association with motor function after stroke. Brain. 2015 Jul;138(Pt 7):1949-60. doi: 10.1093/brain/awv100. Epub 2015 May 1. PMID 25935722
- [Background] Thiel A, Vahdat S. Structural and resting-state brain connectivity of motor networks after stroke. Stroke. 2015 Jan;46(1):296-301. doi: 10.1161/STROKEAHA.114.006307. Epub 2014 Dec 4. No abstract available. PMID 25477218
- [Background] Traversa R, Cicinelli P, Pasqualetti P, Filippi M, Rossini PM. Follow-up of interhemispheric differences of motor evoked potentials from the 'affected' and 'unaffected' hemispheres in human stroke. Brain Res. 1998 Aug 24;803(1-2):1-8. doi: 10.1016/s0006-8993(98)00505-8. PMID 9729235
- [Background] Wang LE, Tittgemeyer M, Imperati D, Diekhoff S, Ameli M, Fink GR, Grefkes C. Degeneration of corpus callosum and recovery of motor function after stroke: a multimodal magnetic resonance imaging study. Hum Brain Mapp. 2012 Dec;33(12):2941-56. doi: 10.1002/hbm.21417. Epub 2011 Oct 22. PMID 22020952
- [Background] Ward NS, Cohen LG. Mechanisms underlying recovery of motor function after stroke. Arch Neurol. 2004 Dec;61(12):1844-8. doi: 10.1001/archneur.61.12.1844. PMID 15596603
- [Background] Weiller C, Ramsay SC, Wise RJ, Friston KJ, Frackowiak RS. Individual patterns of functional reorganization in the human cerebral cortex after capsular infarction. Ann Neurol. 1993 Feb;33(2):181-9. doi: 10.1002/ana.410330208. PMID 8434880
- [Background] Yang M, Yang YR, Li HJ, Lu XS, Shi YM, Liu B, Chen HJ, Teng GJ, Chen R, Herskovits EH. Combining diffusion tensor imaging and gray matter volumetry to investigate motor functioning in chronic stroke. PLoS One. 2015 May 12;10(5):e0125038. doi: 10.1371/journal.pone.0125038. eCollection 2015. PMID 25965398
- [Background] Zheng X, Schlaug G. Structural white matter changes in descending motor tracts correlate with improvements in motor impairment after undergoing a treatment course of tDCS and physical therapy. Front Hum Neurosci. 2015 Apr 30;9:229. doi: 10.3389/fnhum.2015.00229. eCollection 2015. PMID 25983684
- [Derived] Morone G, Capone F, Iosa M, Cruciani A, Paolucci M, Martino Cinnera A, Musumeci G, Brunelli N, Costa C, Paolucci S, Di Lazzaro V. May Dual Transcranial Direct Current Stimulation Enhance the Efficacy of Robot-Assisted Therapy for Promoting Upper Limb Recovery in Chronic Stroke? Neurorehabil Neural Repair. 2022 Dec;36(12):800-809. doi: 10.1177/15459683221138743. PMID 36458455